CLINICAL TRIAL: NCT00805207
Title: Sex Steroids, Sleep, and Metabolic Dysfunction in Women
Acronym: SCOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 07-0692; NIH P50 HD057796
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Obstructive Sleep Apnea; Obesity
Keywords: sleep apnea; obese; Very-low density lipoprotein (VLDL) metabolism; isotope tracer; women
MeSH Terms: conditions — Polycystic Ovary Syndrome; Sleep Apnea, Obstructive; Obesity; Sleep Apnea Syndromes | interventions — Progesterone; Testosterone; Glucocorticoids; Continuous Positive Airway Pressure; Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Progesterone - PCOS (Experimental): Women with obesity and polycystic ovary syndrome
  Interventions: Drug: Progesterone
- Testosterone - premenopausal women (Experimental): Healthy premenopausal women.
  Interventions: Drug: testosterone
- Continuous positive airway pressure (Experimental): Women and men with obesity and obstructive sleep apnea
  Interventions: Device: continuous positive airway pressure
- Glucocorticoid (Experimental): Lean and obese healthy women, and obese men
  Interventions: Drug: glucocorticoid
- Estrogen (Experimental): Postmenopausal women
  Interventions: Drug: Estrogen
- control (Other): Postmenopausal women - tested before and after no treatment. Duration between before and after testing ranged from 31 to 78 days with an average of 46 days between visits
  Interventions: Other: Control
- control - baseline testing only (No Intervention): Healthy men and women
- Progesterone - Postmenopausal women (Experimental): Postmenopausal women
  Interventions: Drug: Progesterone
- Testosterone - Postmenopausal women (Experimental): Postmenopausal women
  Interventions: Drug: testosterone

INTERVENTIONS:
Drug: Progesterone — Micronized progesterone, 100 mg/d vaginally. The intervention lasts 70 days in total and consisted of 14 days on treatment, 14 days off treatment, 14 days on treatment, 14 days off treatment and a final 14 days on treatment. Testing is performed before and at the end of the 70 day intervention.
  Other Names: Endometrin
  Arms: Progesterone - PCOS; Progesterone - Postmenopausal women
Drug: testosterone — Testosterone gel 1250 ug/d applied transdermally for a total of 21 days. Testing is performed before and at the end of the 21 day intervention.
  Other Names: 1% AndroGel
  Arms: Testosterone - Postmenopausal women; Testosterone - premenopausal women
Drug: glucocorticoid — Dexamethasone 0.013 mg/kg fat-free mass daily taken orally for a total of 21 days. Testing is performed before and at the end of the 21 day intervention.
  Arms: Glucocorticoid
Device: continuous positive airway pressure — Breathe through the mask of a continuous positive airway pressure device every night when sleep, for 6 weeks. Testing is performed before and at the end of the 6 week intervention.
  Arms: Continuous positive airway pressure
Drug: Estrogen — Estrogen treatment (100 ug Estradiol daily) administered transdermally by using continuous delivery patches. The intervention lasted 70 days in total and consisted of 14 days on treatment, 14 days off treatment, 14 days on treatment, 14 days off treatment and a final 14 days on treatment.
  Other Names: Estradiol Patch, Mylan Pharmaceuticals Inc.
  Arms: Estrogen
Other: Control — No treatment with studies performed 31 to 72 days apart
  Arms: control

SUMMARY:
Increased plasma triglyceride concentration is a common feature of the metabolic abnormalities associated with obesity and a major risk factor for cardiovascular disease. Obesity is a major risk factor for two conditions that appear to be increasing in prevalence in women: the polycystic ovary syndrome (PCOS) and sleep disordered breathing. PCOS affects 5-8% of women. Sleep disordered breathing affects up to 10% of women. Obstructive sleep apnea (OSA) is the most common cause for sleep disordered breathing and particularly prevalent in obese women with PCOS (~50%). Both PCOS and OSA augment the increase in plasma triglyceride (TG) concentration associated with obesity, and the effects of PCOS and OSA on plasma TG concentration appear to be additive. The mechanisms responsible for the adverse effects on plasma TG metabolism are not known. The primary goal of this project, therefore, is to determine the mechanisms responsible for the increase in plasma TG concentration in obese women with PCOS and OSA. It is our general hypothesis that alterations in the hormonal milieu that are characteristic of these two conditions are, at least in part, responsible for the increase in plasma TG concentration in obese women with the conditions. Furthermore, we hypothesize that the hormonal aberrations characteristic of the two conditions are particularly harmful to obese, compared with lean, women.

The effects of PCOS on skeletal muscle protein metabolism are also not known. However, sex hormones are thought to be important regulators of muscle protein turnover suggesting that muscle protein metabolism is likely to be affected by PCOS. We will examine this by determining the effect of individual sex hormones on muscle protein metabolism and hypothesize that testosterone administration will stimulate muscle protein metabolism while estrogen and progesterone administration will inhibit muscle protein metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-75 years and men 45-75 years
* Healthy lean, overweight and obese women (BMI 18-40 kg/m2) and obese men (BMI 30-40 kg/m2)
* Obese women (BMI 30-40 kg/m2) with OSA or PCOS

Exclusion Criteria:

* Pregnant, lactating, peri- or postmenopausal women will be excluded from the study because of potential confounding influences of these factors and potential ethical concerns (pregnant women)
* Women taking medications known to affect substrate metabolism and those with evidence of significant organ dysfunction (e.g. impaired glucose tolerance, diabetes mellitus, liver disease, hypo- or hyper-thyroidism) other than PCOS and OSA
* Severe hypertriglyceridemia (fasting plasma TG concentration >400 mg/dl)
* Subjects with OSA who have an apnea-hypopnea index (AHI) score >30 (the total number of obstructive events divided by the total hours of sleep) will be excluded and instructed to seek medical care

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Wang X, Magkos F, Patterson BW, Reeds DN, Kampelman J, Mittendorfer B. Low-dose dexamethasone administration for 3 weeks favorably affects plasma HDL concentration and composition but does not affect very low-density lipoprotein kinetics. Eur J Endocrinol. 2012 Aug;167(2):217-23. doi: 10.1530/EJE-12-0180. Epub 2012 May 22. PMID 22619349
- [Result] Wang X, Smith GI, Patterson BW, Reeds DN, Kampelman J, Magkos F, Mittendorfer B. Testosterone increases the muscle protein synthesis rate but does not affect very-low-density lipoprotein metabolism in obese premenopausal women. Am J Physiol Endocrinol Metab. 2012 Mar 15;302(6):E740-6. doi: 10.1152/ajpendo.00533.2011. Epub 2012 Jan 17. PMID 22252942
- [Result] Smith GI, Reeds DN, Okunade AL, Patterson BW, Mittendorfer B. Systemic delivery of estradiol, but not testosterone or progesterone, alters very low density lipoprotein-triglyceride kinetics in postmenopausal women. J Clin Endocrinol Metab. 2014 Jul;99(7):E1306-10. doi: 10.1210/jc.2013-4470. Epub 2014 Apr 2. PMID 24694337
- [Result] Smith GI, Yoshino J, Reeds DN, Bradley D, Burrows RE, Heisey HD, Moseley AC, Mittendorfer B. Testosterone and progesterone, but not estradiol, stimulate muscle protein synthesis in postmenopausal women. J Clin Endocrinol Metab. 2014 Jan;99(1):256-65. doi: 10.1210/jc.2013-2835. Epub 2013 Dec 20. PMID 24203065

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Positive Airway Pressure: Obese women and men with obstructive sleep apnea
  continuous positive airway pressure: Breathe through the mask of a continuous positive airway pressure device every night when sleep, for 6 weeks
- Glucocorticoid: Lean and obese healthy women, and obese men
  glucocorticoid: Dexamethasone 0.013 mg/kg fat-free mass daily, 21 days
- Estrogen: Postmenopausal women
  Estrogens: Estrogen treatment (100 ug Estradiol daily) administered 14 days followed by 14 days without treatment. Repeat this cycle 3 times.
- Control - Baseline Testing Only: Baseline testing only in pre- and postmenopausal women
Period: Overall Study
Arm/Group | Progesterone - PCOS | Progesterone - Postmenopausal Women | Testosterone - Premenopausal Women | Testosterone - Postmenopausal Women | Continuous Positive Airway Pressure | Glucocorticoid | Estrogen | Control | Control - Baseline Testing Only
Started | 1 | 9 | 12 | 6 | 3 | 12 | 6 | 6 | 6
Completed | 1 | 7 | 11 | 6 | 2 | 9 | 6 | 6 | 6
Not Completed | 0 | 2 | 1 | 0 | 1 | 3 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Testosterone - Premenopausal Women: Healthy, premenopausal women
  Testosterone gel 1250 ug/d applied transdermally for a total of 21 days. Testing is performed before and at the end of the 21 day intervention
- Testosterone - Postmenopausal Women: Postmenopausal women
  Testosterone gel 1250 ug/d applied transdermally for a total of 21 days. Testing is performed before and at the end of the 21 day intervention.
- Progesterone - PCOS: Women with obesity and polycystic ovary syndrome
  Micronized progesterone, 100 mg/d vaginally. The intervention lasts 70 days in total and consisted of 14 days on treatment, 14 days off treatment, 14 days on treatment, 14 days off treatment and a final 14 days on treatment. Testing is performed before and at the end of the 70 day intervention.
- Progesterone - Postmenopausal Women: Postmenopausal women
  Micronized progesterone, 100 mg/d vaginally. The intervention lasts 70 days in total and consisted of 14 days on treatment, 14 days off treatment, 14 days on treatment, 14 days off treatment and a final 14 days on treatment. Testing is performed before and at the end of the 70 day intervention.
- Continuous Positive Airway Pressure: Women and men with obesity and obstructive sleep apnea
  continuous positive airway pressure: Breathe through the mask of a continuous positive airway pressure device every night when sleep, for 6 weeks
- Control: Postmenopausal women
  Tested before and after no treatment. Duration between before and after testing ranged from 31 to 78 days with an average of 46 days between visits
- Control - Baseline Testing Only: Healthy men and women
  Baseline testing only
- Total: Total of all reporting groups
Arm/Group | Testosterone - Premenopausal Women | Testosterone - Postmenopausal Women | Progesterone - PCOS | Progesterone - Postmenopausal Women | Continuous Positive Airway Pressure | Glucocorticoid | Estrogen | Control | Control - Baseline Testing Only | Total
Number analyzed (Participants) | 12 | 6 | 1 | 9 | 3 | 12 | 6 | 6 | 6 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (8) | 57 (6) | 22 (0) | 63 (7) | 62 (12) | 38 (13) | 59 (10) | 64 (6) | 41 (15) | 49 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 1 | 9 | 2 | 9 | 6 | 6 | 5 | 56
  Male | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 2 | 0 | 2 | 2 | 3 | 0 | 0 | 3 | 19
  White | 5 | 4 | 1 | 7 | 1 | 8 | 6 | 6 | 3 | 41
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 1 | 9 | 3 | 12 | 6 | 6 | 6 | 61

OUTCOME MEASURES:

1. Primary Outcome: Very-Low Density Lipoprotein-Triglyceride (VLDL-TG) Secretion Rate
Description: VLDL was isolated from plasma by ultracentrifugation with the tracer-to-tracee (TTR) of free glycerol in plasma and glycerol in VLDL-TG determined by gas chromatography-mass spectrometry. The fractional turnover rates of VLDL-TG was determined by fitting the glycerol TTR time courses in plasma and in VLDL-TG to a multicompartmental model. The hepatic (liver) secretion rates of VLDL-TG was calculated by multiplying the fractional turnover rates of VLDL-TG by the of VLDL-TG concentration.
Time Frame: Before and at the end of interventions
Population: Not included in final analysis:
  Withdrawn/withdrew= Testosterone premenopausal women x 1; Progesterone postmenopausal women x 2; Glucocorticoid x 3.
  VLDL-TG fractional turnover rate was 3 Standard Deviations from the mean = Testosterone - premenopausal women x 1.
  Undetectable VLDL-TG concentration = Progesterone - Postmenopausal women x 1.
Measure: Mean (Standard Deviation); unit: umol/min/L plasma
Groups:
- Testosterone - Premenopausal Women: Healthy, premenopausal women.
  Testosterone gel 1250 ug/d applied transdermally for a total of 21 days. Testing is performed before and at the end of the 21 day intervention.
Arm/Group | Testosterone - Premenopausal Women | Testosterone - Postmenopausal Women | Progesterone - PCOS | Progesterone - Postmenopausal Women | Continuous Positive Airway Pressure | Glucocorticoid | Estrogen | Control | Control - Baseline Testing Only
Number analyzed (Participants) | 10 | 6 | 1 | 6 | 2 | 9 | 6 | 6 | 6
umol/min/L plasma
  Before | 3.13 (2.11) | 2.03 (0.35) | 4.66 | 3.36 (1.65) | 2.87 (0.03) | 3.80 (1.52) | 2.87 (0.86) | 2.47 (0.85) | 3.53 (2.88)
  After: number analyzed (Participants) | 10 | 6 | 1 | 6 | 2 | 9 | 6 | 6 | 0
  After | 3.00 (1.58) | 2.11 (0.80) | 7.77 | 3.24 (1.55) | 3.94 (0.42) | 3.42 (2.01) | 2.94 (1.40) | 2.57 (1.26) |
Statistical Analysis 1: Comparison: Testosterone - Premenopausal Women; Test type: Other; p = 0.85, t-test, 2 sided
Statistical Analysis 2: Comparison: Glucocorticoid; Test type: Other; p = 0.70, t-test, 2 sided
Statistical Analysis 3: Comparison: Testosterone - Postmenopausal Women vs Progesterone - Postmenopausal Women vs Estrogen vs Control; Test type: Other; p = 0.88, ANOVA — P-value is the main effect of treatment (i.e., Before vs. After) from ANOVA; VLDL-TG secretion rates were skewed and log transformed prior to performing ANOVA
Statistical Analysis 4: Comparison: Testosterone - Postmenopausal Women vs Progesterone - Postmenopausal Women vs Estrogen vs Control; Test type: Other; p = 0.26, ANOVA — P-value is the main effect of group (i.e., Testosterone, Progesterone, Estrogen and Control) from ANOVA; VLDL-TG secretion rates were skewed and log transformed prior to performing ANOVA
Statistical Analysis 5: Comparison: Testosterone - Postmenopausal Women vs Progesterone - Postmenopausal Women vs Estrogen vs Control; Test type: Other; p = 0.98, ANOVA — P value is the group by treatment interaction from the ANOVA; VLDL-TG secretion rates were skewed and log transformed prior to performing ANOVA

2. Secondary Outcome: Very-Low Density Lipoprotein-Triglyceride (VLDL-TG) Concentration
Description: VLDL was isolated from plasma by ultracentrifugation with VLDL-TG concentration measured by using a colorimetric enzymatic kit (Sigma-Aldrich, St. Louis, MO).
Time Frame: Before and at the end of the interventions
Population: Not included in final analysis:
  Withdrawn/withdrew = Testosterone premenopausal women x 1; Progesterone postmenopausal women x 2; Glucocorticoid x 3.
  VLDL-TG fractional turnover rate was 3 Standard Deviations from the mean = Testosterone - premenopausal women x 1.
  Undetectable VLDL-TG concentration = Progesterone - Postmenopausal women x 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Testosterone - Premenopausal Women | Testosterone - Postmenopausal Women | Progesterone - PCOS | Progesterone - Postmenopausal Women | Continuous Positive Airway Pressure | Glucocorticoid | Estrogen | Control | Control - Baseline Testing Only
Number analyzed (Participants) | 10 | 6 | 1 | 6 | 2 | 9 | 6 | 6 | 6
mmol/L
  Before | 0.31 (0.29) | 0.18 (0.09) | 0.75 | 0.42 (0.18) | 0.50 (0.06) | 0.35 (0.16) | 0.50 (0.28) | 0.30 (0.15) | 0.32 (0.17)
  After: number analyzed (Participants) | 10 | 6 | 1 | 6 | 2 | 9 | 6 | 6 | 0
  After | 0.40 (0.50) | 0.18 (0.10) | 1.03 | 0.44 (0.36) | 0.64 (0.18) | 0.33 (0.22) | 0.35 (0.22) | 0.28 (0.16) |
Statistical Analysis 1: Comparison: Testosterone - Premenopausal Women; Test type: Other; p = 0.31, t-test, 2 sided
Statistical Analysis 2: Comparison: Glucocorticoid; Test type: Other; p = 0.82, t-test, 2 sided
Statistical Analysis 3: Comparison: Estrogen vs Control; Test type: Other; p < 0.05, ANCOVA
Statistical Analysis 4: Comparison: Progesterone - Postmenopausal Women vs Control; Test type: Other; p = 0.87, ANCOVA
Statistical Analysis 5: Comparison: Testosterone - Postmenopausal Women vs Control; Test type: Other; p = 0.57, ANCOVA

3. Secondary Outcome: VLDL-TG Plasma Clearance Rate (Means)
Description: VLDL was isolated from plasma by ultracentrifugation with the tracer-to-tracee (TTR) of free glycerol in plasma and glycerol in VLDL-TG determined by gas chromatography-mass spectrometry. The fractional turnover rates of VLDL-TG was determined by fitting the glycerol TTR time courses in plasma and in VLDL-TG to a multicompartmental model. The plasma clearance rate of VLDL-TG was calculated by dividing the VLDL-TG secretion rate by the VLDL-TG concentration.
Time Frame: Before and at the end of the interventions
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Groups:
- Testosterone - Premenopausal Women: Healthy premenopausal women.
  Testosterone gel 1250 ug/d applied transdermally for a total of 21 days. Testing is performed before and at the end of the 21 day intervention.
- Control: Postmenopausal women
  Postmenopausal women - tested before and after no treatment. Duration between before and after testing ranged from 31 to 78 days with an average of 46 days between visits
Arm/Group | Testosterone - Premenopausal Women | Testosterone - Postmenopausal Women | Progesterone - PCOS | Progesterone - Postmenopausal Women | Continuous Positive Airway Pressure | Glucocorticoid | Estrogen | Control | Control - Baseline Testing Only
Number analyzed (Participants) | 10 | 6 | 1 | 6 | 3 | 9 | 6 | 6 | 6
mL/min
  Before: number analyzed (Participants) | 10 | 6 | 1 | 6 | 2 | 9 | 6 | 6 | 4
  Before | 42.2 (16.3) | 35.1 (16.5) | 20.3 | 21.2 (7.5) | 19.1 (2.7) | 33.8 (11.3) | 17.4 (6.7) | 22.6 (9.0) | 33.1 (13.1)
  After: number analyzed (Participants) | 10 | 6 | 1 | 6 | 2 | 9 | 6 | 6 | 0
  After | 58.1 (51.6) | 34.5 (15.8) | 24.6 | 24.9 (15.3) | 20.8 (2.8) | 34.3 (21.9) | 25.1 (6.1) | 23.3 (5.0) |
Statistical Analysis 1: Comparison: Glucocorticoid; Test type: Other; p = 0.94, t-test, 2 sided
Statistical Analysis 2: Comparison: Estrogen vs Control; Test type: Other; p < 0.05, ANCOVA
Statistical Analysis 3: Comparison: Progesterone - Postmenopausal Women vs Control; Test type: Other; p = 0.53, ANCOVA
Statistical Analysis 4: Comparison: Testosterone - Postmenopausal Women vs Control; Test type: Other; p = 0.23, ANCOVA

4. Secondary Outcome: VLDL-TG Plasma Clearance Rate (Medians)
Description: as for outcome 3
Time Frame: Before and at the end of the interventions
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | Testosterone - Premenopausal Women | Testosterone - Postmenopausal Women | Progesterone - PCOS | Progesterone - Postmenopausal Women | Continuous Positive Airway Pressure | Glucocorticoid | Estrogen | Control | Control - Baseline Testing Only
Number analyzed (Participants) | 10 | 6 | 1 | 6 | 3 | 9 | 6 | 6 | 6
mL/min
  Before: number analyzed (Participants) | 10 | 6 | 1 | 6 | 3 | 9 | 6 | 6 | 4
  Before | 40.6 [33.8 to 52.9] | 32.1 [23.1 to 47.8] | 20.3 | 20.8 [15.4 to 25.4] | 19.1 [18.1 to 20.1] | 35.8 [29.6 to 40.5] | 14.4 [12.7 to 20.5] | 19.6 [16.6 to 26.8] | 33.4 [22.8 to 43.7]
  After: number analyzed (Participants) | 10 | 6 | 1 | 6 | 3 | 9 | 6 | 6 | 0
  After | 43.6 [19.4 to 63.5] | 32.7 [24.4 to 48.1] | 20.3 | 22.8 [15.7 to 34.3] | 20.8 [19.9 to 21.8] | 27.4 [21.5 to 38.7] | 24.2 [22.0 to 29.1] | 22.3 [19.0 to 26.9] |
Statistical Analysis 1: Comparison: Testosterone - Premenopausal Women; Test type: Other; p = 0.80, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Basal, Postabsorptive Fractional Synthesis Rates of Muscle Protein Synthesis
Description: The fractional synthesis rate (FSR) of muscle protein synthesis was determined by assessing the incorporation of [5,5,5-2H3]leucine into muscle proteins. [5,5,5-2H3]leucine was infused for 5 hours with muscle biopsies obtained from the vastus lateralis muscle in the thigh 2 and 5 hours. The leucine tracer-to-tracee ratio (TTR) in muscle protein and the muscle free leucine pool was determined by gas chromatography-mass spectrometry (GCMS) and the FSR of muscle proteins calculated using a standard precursor-product model.
  The FSR was calculated as %/h, which reflects the percent of all proteins in the muscle that were synthesized (made) per hour.
Time Frame: Before and at the end of the intervention
Population: Not included in final analysis:
  Withdrawn/withdrew = Testosterone premenopausal women x 1; Progesterone postmenopausal women x 2; Glucocorticoid x 3.
  Muscle not obtained = Testosterone - premenopausal women x 1; Progesterone postmenopausal women x 1; CPAP x 3; Glucocorticoid x 6; Control - baseline testing only x 6.
Measure: Mean (Standard Deviation); unit: %/h
Arm/Group | Testosterone - Premenopausal Women | Testosterone - Postmenopausal Women | Progesterone - PCOS | Progesterone - Postmenopausal Women | Continuous Positive Airway Pressure | Glucocorticoid | Estrogen | Control | Control - Baseline Testing Only
Number analyzed (Participants) | 10 | 6 | 1 | 6 | 0 | 3 | 6 | 6 | 0
%/h
  Before | 0.064 (0.023) | 0.056 (0.007) | 0.049 | 0.054 (0.12) |  | 0.059 (0.007) | 0.063 (0.016) | 0.064 (0.012) |
  After | 0.092 (0.024) | 0.079 (0.030) | 0.083 | 0.085 (0.018) |  | 0.061 (0.037) | 0.063 (0.026) | 0.067 (0.011) |
Statistical Analysis 1: Comparison: Testosterone - Premenopausal Women; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Testosterone - Postmenopausal Women vs Progesterone - Postmenopausal Women vs Estrogen vs Control; Test type: Other; p < 0.01, ANOVA — P-value is the main effect of treatment (i.e., Before vs. After) from ANOVA
Statistical Analysis 3: Comparison: Testosterone - Postmenopausal Women vs Progesterone - Postmenopausal Women vs Estrogen vs Control; Test type: Other; p = 0.96, ANOVA — P-value is the main effect of group (i.e., Testosterone, Progesterone, Estrogen and Control) from ANOVA
Statistical Analysis 4: Comparison: Testosterone - Postmenopausal Women vs Progesterone - Postmenopausal Women vs Estrogen vs Control; Test type: Other; p < 0.05, ANOVA — P value is the group by treatment interaction from the ANOVA
Statistical Analysis 5: Comparison: Testosterone - Postmenopausal Women; Test type: Other; p < 0.01, Tukey test
Statistical Analysis 6: Comparison: Progesterone - Postmenopausal Women; Test type: Other; p < 0.01, Tukey test
Statistical Analysis 7: Comparison: Estrogen; Test type: Other; p > 0.10, Tukey test
Statistical Analysis 8: Comparison: Control; Test type: Other; p > 0.10, Tukey test

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the following periods; Estrogen = 70 days (consisted of 14 days on treatment, 14 days off treatment, 14 days on treatment, 14 days off treatment and a final 14 days on treatment.); Testosterone = 21 days; continuous positive airway pressure = 6 weeks; Dexamethasone = 21 days; Progesterone = 70 days (consisted of 14 days on, 14 days off, 14 days on, 14 days off and a final 14 days on treatment); Control (no treatment) = 31 to 72 days between testing visits.
Groups:
- Continuous Positive Airway Pressure: Obese women and men with obstructive sleep apnea
  Breathe through the mask of a continuous positive airway pressure device every night when sleep, for 6 weeks. Testing is performed before and at the end of the 6 week intervention.
Arm/Group | Testosterone - Premenopausal Women | Testosterone - Postmenopausal Women | Progesterone - PCOS | Progesterone - Postmenopausal Women | Continuous Positive Airway Pressure | Glucocorticoid | Estrogen | Control | Control - Baseline Testing Only
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/1 | 0/9 | 0/3 | 0/12 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/1 | 0/9 | 0/3 | 0/12 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/3 | 3/9 | 0/3 | 0/12 | 1/6 | 0/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone - Premenopausal Women (N=12) | Testosterone - Postmenopausal Women (N=6) | Progesterone - PCOS (N=3) | Progesterone - Postmenopausal Women (N=9) | Continuous Positive Airway Pressure (N=3) | Glucocorticoid (N=12) | Estrogen (N=6) | Control (N=6) | Control - Baseline Testing Only (N=6)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — One subject reported that she had more acne that usual while taking estrogen
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — One subject reported that she had a small amount of vaginal discharge while taking estrogen
Itchiness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — On subject reported her ankles were itchy while on progesterone
Shaking (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — One subject in the progesterone group contacted us saying that she was shaking violently while not on treatment. Unrelated to treatment was probably due to a viral infection.
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — One subject in the progesterone group contacted us saying that she was vomiting while not on treatment. Unrelated to treatment was probably due to a viral infection.
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — One subject in the progesterone group contacted us saying that she had diarrhea while not on treatment. Unrelated to treatment was probably due to a viral infection.
Broken ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Subject in Progesterone group broke her ankle while on treatment but unrelated to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No